CLINICAL TRIAL: NCT04471870
Title: Multicentre Observational, Prospective Cohort Study Including Patients With Acute Coronary Syndromes Undergoing Percutaneous Coronary Intervention Who Receive Cangrelor i.v. Transitioning to Clopidogrel, Prasugrel or Ticagrelor Per os
Brief Title: ARCANGELO (itAlian pRospective Study on CANGrELOr)
Acronym: ARCANGELO
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: DFIDM-1801
Record Dates: First submitted 2020-07-06; First posted 2020-07-15 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome
Keywords: Real-word; ACS; PCI
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Sponsor implemented a post-authorisation safety study (PASS), category 3, focused in Acute Coronary Syndrome, in order to collect information about the safety of cangrelor in the real clinical practice, evaluating the safety of the transition to all the oral P2Y12 inhibitors (cangrelor, ticagrelor and prasugrel).

ELIGIBILITY:
Inclusion Criteria:

1. Patients' written informed and privacy consent obtained before or at the end of the PCI procedure according to patients' condition but in any case, prior to collection of any study-related data;
2. Male or female patients aged ≥ 18 years;
3. Patients with acute coronary syndromes undergoing PCI;
4. Patients who are planned to be treated with cangrelor, or who have received treatment with cangrelor.

Exclusion Criteria:

1. Patients with active bleeding or increased risk of bleeding, because of impaired haemostasis and/or irreversible coagulation disorders or due to recent major surgery/trauma or uncontrolled severe hypertension;
2. Patients with history of stroke or transient ischaemic attack (TIA);
3. Patients with hypersensitivity to the active substance (cangrelor) or to any of its excipients;
4. Known pregnancy or breast-feeding female patients;
5. Patients with stable angina (SA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndromes undergoing percutaneous coronary intervention who receive cangrelor i.v. according to the clinical practice
Sampling Method: Probability Sample
Enrollment: 1005 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence of any haemorrages according to BARC (Bleeding Academic Research Consortium) criteria | 30 days post-PCI
  The incidence will be calculated as the ratio between the number of patients experiencing at least one event during the 30-day observation period over the total number of evaluable patients.

SECONDARY OUTCOMES:
Incidence of type 1-2 (mild) bleedings, according to the Bleeding Academic Research Consortium [BARC] criteria | 48 hours after PCI
  The incidence will be calculated as the ratio between the number of evaluable patients who experience at least one event and the total number of evaluable patients
Incidence of type 1-2 (mild) bleedings, according to the Bleeding Academic Research Consortium [BARC] criteria | 30 days after PCI
  The incidence will be calculated as the ratio between the number of evaluable patients who experience at least one event and the total number of evaluable patientsConsortium [BARC]
Incidence of type 3-5 (moderate severe) bleedings, according to the Bleeding Academic Research Consortium [BARC] criteria | 48 hours after PCI
  The incidence will be calculated as the ratio between the number of evaluable patients who experience at least one event and the total number of evaluable patientsConsortium [BARC]
Incidence of type 3-5 (moderate severe) bleedings, according to the Bleeding Academic Research Consortium [BARC] criteria | 30 days after PCI
  The incidence will be calculated as the ratio between the number of evaluable patients who experience at least one event and the total number of evaluable patientsConsortium [BARC] bleedings, according to the Bleeding Academic Research Consortium [BARC]
Incidence of major adverse cardiac events (MACE) | 48 hours after PCI
  The incidence will be calculated as the ratio between the number of evaluable patients who experience at least one event and the total number of evaluable patients. MACE will comprise any of the following events: death, myocardial infarction (MI), ischemia-driven revascularisation (IDR) and stent thrombosis (ST).
Incidence of major adverse cardiac events (MACE) | 30 days after PCI
  The incidence will be calculated as the ratio between the number of evaluable patients who experience at least one event and the total number of evaluable patients. MACE will comprise any of the following events: death, myocardial infarction (MI), ischemia-driven revascularisation (IDR) and stent thrombosis (ST).
To describe the type of oral platelet P2Y12 receptor (prasugrel/ticagrelor/clopidogrel) | 30 days after PCI
  It will be calculated the proportion of patients receiving an oral platelet P2Y12 receptor in terms of type (prasugrel/ticagrelor/clopidogrel) and timing of administration
To describe the use of glycoprotein IIb/IIIa (GPIIb/IIIa) inhibitors | 30 days after PCI
  It will be calculated the proportion of patients receiving GPIIb/IIIa inhibitors

CONTACTS AND LOCATIONS:
Locations (30):
- Italy (30):
  - A.O.U. Riuniti, Ancona
  - Ospedale San Donato, Arezzo
  - A.O.U. Consorziale Policlinico, Bari
  - Ospedale San Bassiano, Bassano del Grappa
  - Azienda Ospedaliera San Pio, Benevento
  - Ospedale Maggiore, Bologna
  - Fondazione Poliambulanza, Brescia
  - A.O. Sant'Anna e San Sebastiano, Caserta
  - A.O.U. Policlinico-Vittorio Emanuele P.O. Ferrarotto, Catania
  - Ospedale SS Annunziata, Cosenza
  - ASO Santa Croce e Carle, Cuneo
  - A.O.U. Careggi, Florence
  - Ospedale Fabrizio Spaziani, Frosinone
  - Ospedale S. Andrea, La Spezia
  - Ospedale Santa Maria Goretti, Latina
  - Fondazione Toscana "G. Monasterio" Ospedale del Cuore G. Pasquinucci, Massa
  - Centro Cardiologico Monzino, Milan
  - A.O.R.N. A. Cardarelli, Napoli
  - A.O.U. Federico II, Napoli
  - A.O. Padova, Padua
  - Policlinico San Matteo, Pavia
  - Ospedale degli Infermi, Rivoli
  - San Camillo Forlanini, Roma
  - Aurelia Hospital, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - A.O.U. Sassari, Sassari
  - Ospedale Umberto I, Syracuse
  - A.O. Mauriziano, Torino
  - Ospedale Santa Chiara, Trento
  - Ospedale Ca' Foncello, Treviso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capranzano P, Calabro P, Musumeci G, Mario CD, Chirillo F, Rolfo C, Menozzi A, Menichelli M, Maffeo D, Talanas G, Ferlini M, Contarini M, Lanzilotti V, De Luca L. Use of Cangrelor in Older Patients: Findings from the itAlian pRospective Study on CANGrELOr Study. Am J Cardiol. 2025 Apr 1;240:31-37. doi: 10.1016/j.amjcard.2024.12.021. Epub 2024 Dec 21. PMID 39716523